CLINICAL TRIAL: NCT02820350
Title: A Multi-Center, Pilot Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device (SCD) in Pediatric Patients With Acute Kidney Injury (AKI)
Brief Title: Safety and Efficacy of a Selective Cytopheretic Device (SCD) in Pediatric Patients With Acute Kidney Injury (AKI).
Acronym: SCD-PED-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CytoPherx, Inc (Industry)
Collaborators: Innovative BioTherapies (IBT) (Industry); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCD-PED-01; FD005092-01 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2016-06-07; First posted 2016-06-30 (Estimated); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute Renal Failure; Acute kidney injury; Continuous Renal Replacement Therapy; Selective cytopheretic device; Pediatric
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other): Treatment arm only
  Interventions: Device: SCD-F40

INTERVENTIONS:
Device: SCD-F40 — CRRT with SCD
  Other Names: Selective Cytopheretic Device (SCD)

SUMMARY:
The SCD (Selective Cytopheretic Device) is an extracorporeal device used as an adjunct to renal replacement therapy (RRT) to improve the outcomes of pediatric patients with acute kidney injury (AKI). Funding Source - FDA OOPD (SCD-PED-01)

DETAILED DESCRIPTION:
The selective cytopheretic device (SCD) is comprised of tubing, connectors and a hemofilter cartridge. The device is connected in series to commercially available Continuous Renal Replacement Therapy (CRRT) devices. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and it is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.

ELIGIBILITY:
Inclusion Criteria:

1. A patient, or legal representative, has signed a written informed consent form.
2. Must be receiving medical care in an intensive care unit (e.g., ICU, MICU, SICU, CTICU, Trauma).
3. Age less than 22 years.
4. Females of child bearing potential who are not pregnant (confirmed by a negative serum pregnancy test) and not lactating if recently post-partum.
5. Intent to deliver full supportive care through aggressive management utilizing all available therapies for a minimum of 96 hours.
6. Clinical diagnosis of AKI due to etiologies requiring CRRT (see Appendix B). AKI is defined as acute kidney injury with any one of the following:

   * Increase in SCr by ≥0.3 mg/dL (≥26.5 μmol/L) within 48 hours or;
   * Increase in SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days or;
   * Urine volume <0.5ml/kg/h for 6 hours
7. At least one non-renal organ failure (defined as receiving mechanical ventilation or at least one vasoactive medication to treat hypotension) OR presence (proven or suspected) of sepsis. (Appendix C).

Exclusion Criteria:

1. Irreversible brain damage based on available historical and clinical information.
2. Presence of any organ transplant at any time.
3. Acute or chronic use of circulatory support device such as LVADs, RVADs, BIVADs, ECMO(a).
4. Presence of preexisting advanced chronic renal failure (i.e., ESRD) requiring CRRT prior to this episode of AKI.
5. AKI occurring in the setting of burns, obstructive uropathy, allergic interstitial nephritis, acute or rapidly progressive glomerulonephritis, vasculitis, hemolytic-uremic syndrome(b), thrombotic thrombocytopenic purpura (TTP), malignant hypertension, scleroderma renal crisis, atheroembolism, functional or surgical nephrectomy, hepatorenal syndrome, cyclosporine, or tacrolimus nephrotoxicity
6. Received >12hrs of CRRT during this hospital admission or prior to transfer from an outside hospital.
7. Received >1 hemodialysis treatment during this hospital admission or prior to transfer from an outside hospital.
8. Hospitalization >14 days during this hospital admission and or prior to transfer from an outside hospital.
9. Metastatic malignancy which is actively being treated or may be treated by chemotherapy or radiation during the subsequent three-month period after study therapy.
10. Chronic immunosuppression.
11. HIV or AIDS.
12. Severe liver failure(c).
13. Current Do Not Attempt Resuscitation (DNAR), Allow Natural Death (AND), or withdrawal of care status, or anticipated change in status within the next 7 days.
14. Patient is moribund or chronically debilitated for whom full supportive care is not indicated.
15. Patient not expected to survive 28 days because of an irreversible medical condition. (This is not restrictive to AKI, and may include situations such as the presence of irreversible brain damage, untreatable malignancy, inoperable life threatening condition, or any condition to which therapy is regarded as futile by the PI.)
16. Any medical condition that the Investigator thinks may interfere with the study objectives.
17. Physician refusal.
18. Dry weight of <20kg(d).
19. Platelet count <30,000/mm3 at time of screening(e).
20. Concurrent enrollment in another interventional clinical trial. Patients enrolled in clinical trials where only measurements and/or samples are taken (NO TEST DEVICE OR TEST DRUG USED) are allowed to participate.
21. Use of any other Investigational drug or device within the previous 30 days.

    1. ECMO was subsequently removed as an exclusion. Two patients in the study received ECMO.
    2. Hemolytic uremic syndrome subsequently removed as an exclusion. One patient in the study had HUS.
    3. Severe liver failure was change to severe chronic liver failure during the study course.
    4. The lower weight limit threshold was decreased to 15 kg after consultation and approval from the US FDA.
    5. The thrombocytopenia exclusion removed after no observed occurrences in the first five subjects.

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2016-12-04 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein SL, Askenazi DJ, Basu RK, Selewski DT, Paden ML, Krallman KA, Kirby CL, Mottes TA, Terrell T, Humes HD. Use of the Selective Cytopheretic Device in Critically Ill Children. Kidney Int Rep. 2020 Dec 19;6(3):775-784. doi: 10.1016/j.ekir.2020.12.010. eCollection 2021 Mar. PMID 33732992
- See also: Digital Object Identifier) — http://doi.org/10.1016/j.ekir.2020.12.010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 subjects have been consented for this trial. 16 of the nineteen went on to receive the SCD device.
Groups:
- CRRT + SCD: The Selective Cytopheretic Device (SCD) is comprised of tubing, connectors, and a synthetic membrane cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemoﬁlter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and it is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.
Period: Overall Study
Arm/Group | CRRT + SCD
Started | 19
Completed | 12
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | CRRT + SCD
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 12.3 [4.3 to 20.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Adverse events related to device treatment occurring during and 60 days post treatment initiation
Time Frame: 60 days post treatment initiation
Population: Adverse events related to SCD treatment up to 60 days following treatment initiation
Measure: Number; unit: adverse event
Arm/Group | Treatment
Number analyzed (Participants) | 16
adverse event | 0

2. Secondary Outcome: All Cause Mortality Through 60 Days Post-randomization.
Description: The effect of SCD treatment on all cause mortality through 60 days post-randomization.
Time Frame: Day 60
Population: Outcome data is reported for those subjects in which the calcium levels were maintained in the protocol's recommended range (≤0.4 mmol/L) for greater or equal to 90% of the therapy time.
Measure: Count of Participants; unit: Participants
Groups:
- CRRT + SCD: SCD treated group
Arm/Group | CRRT + SCD
Number analyzed (Participants) | 16
Participants
  Survival | 12
  Non-survival | 4

3. Secondary Outcome: Mortality at Day 28
Description: Mortality at day 28 following treatment
Time Frame: Day 28 following treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- CRRT + SCD: SCD Treatment
Arm/Group | CRRT + SCD
Number analyzed (Participants) | 16
Participants
  Survival | 16
  Non survival | 0

4. Secondary Outcome: The Effect of SCD Treatment on Renal Replacement Therapy Dependency at Day 60.
Description: RRT dependency at day 60 is defined as patient not receiving any form of intermittent or continuous renal replacement therapy at 60 days post enrollment in the study with no plans for additional intermittent or continuous renal replacement therapy.
Time Frame: 60 days
Population: Survivors at day 60
Measure: Count of Participants; unit: Participants
Arm/Group | CRRT + SCD
Number analyzed (Participants) | 12
Participants
  No dialysis dependency | 12
  Dialysis dependency | 0

ADVERSE EVENTS:
Time Frame: During and 60 Days Post Treatment Initiation.
Arm/Group | CRRT + SCD
All-Cause Mortality (participants affected / at risk) | 4/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRRT + SCD (N=16)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4)
Pneumoperitoneum (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Cerebral Hemorrhage (Nervous system disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Vascular Graft Occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRRT + SCD (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) — Thrombocytopenia, Thrombocytosis and Heparin-induced thrombocytopenia
Tachycardia (Cardiac disorders) | 3 (3) — Tachycardia
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) — Hyperglycemia, Hypokalemia
Hypertension (Vascular disorders) | 7 (7) — Hypertension, Hypotension, Pulmonary hemorrhage
Post procedure pneumonia (Infections and infestations) | 1 (1) — Post procedure pneumonia (hospital-acquired)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) — Cerebral hemorrhage
Hypothermia (General disorders) | 5 (5) — Hypothermia, Pyrexia
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) — Pneumoperitoneum
Subcutaneous emphysema (Injury, poisoning and procedural complications) | 1 (1) — Subcutaneous emphysema
Intensive care unit delirium (Psychiatric disorders) | 1 (1) — Intensive care unit delirium
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Acute respiratory failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT02820350/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT02820350/ICF_001.pdf